CLINICAL TRIAL: NCT01448174
Title: Salusin-alpha - a New Factor in the Pathogenesis of Lipid Abnormalities in Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Alicja E. Grzegorzewska, Full Professor, Poznan University of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: ALGN-001
Record Dates: First submitted 2011-10-05; First posted 2011-10-07 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Renal Failure Chronic Requiring Hemodialysis; Metabolic Syndrome; Diabetes Mellitus Type 2; Hyperlipidemia
Keywords: salusin-alpha; atorvastatin; CD36; Hemodialysis
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus, Type 2; Hyperlipidemias | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- atorvastatin (Active Comparator): The prospective, randomized, double-blind, placebo-controlled study:
  * will be preceded by one month non-pharmacological treatment of hyperlipidemia (prerandomization phase)
  * 130 hyperlipidemic hemodialysis (HD) patients will be randomly assigned to receive blinded study drug: 65 patients will be allocated to start with atorvastatin and 65 patients - with placebo.
  Atorvastatin will be administered and monitored according to the K/DOQI guidelines (2003).
  The prospective, observational study:
  - 35 hyperlipidemic patients will be followed for 30 weeks on the prescribed non-pharmacological treatment of hyperlipidemia
  Interventions: Drug: Atorvastatin
- Lifestyle counseling (No Intervention): Protocol of the prospective study in obese persons:
  * after taking the anthropometric measurements and collecting a blood sample, the start of weight lowering therapy with a prescribed diet and planned physical activity
  * follow-up for 30 weeks (measurement of body weight every week).
- The controls (healthy volunteers) (No Intervention)

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin (10 - 80 mg/day) will be administered orally in the one evening dose in the case of strict indications for such a treatment. Before starting atorvastatin, serum lipid profile will be examined two times, and when both results are abnormal the treatment is started. Duration of administration:
  * atorvastatin 12 weeks, 6 weeks washout, placebo 12 weeks or
  * placebo 12 weeks,6 weeks washout,atorvastatin 12 weeks.
  Other Names: ATC: C 10 AA 05
  Arms: atorvastatin

SUMMARY:
Hyperlipidemia and atherosclerosis lead to cardiovascular diseases and are an indirect cause of increased death rate in the general population. This association is still more evident in specific subpopulations, like patients with advanced chronic kidney disease (CKD), especially hemodialysis (HD) patients, due to a higher prevalence of lipid disturbances and atherosclerosis compared to the general population. Cardiovascular events in CKD patients are frequently associated with traditional risk factors, including diabetes, male sex, hypertension, dyslipidemia and advanced age. However, these factors failed to fully account for the increased risk of cardiovascular events in CKD. The efforts are made to identify new risk factors that contribute to the development of atherosclerosis and participate in causes of cardiovascular death. In 2003, there were identified peptides designated salusin-alpha and salusin-beta. Development of atherosclerosis may be suppressed by salusin-alpha. Salusin-alpha may have a lipid lowering effect, similar to that of statins.

The purpose of this study is to investigate whether 1) salusin-alpha is associated with lipid metabolism of HD patients (without or with metabolic syndrome or type 2 diabetes mellitus), similarly or not like in healthy or obese subjects; 2) treatment with atorvastatin and its effects are associated with changes in plasma salusin-alpha concentration, if so - whether it is dependent on the direct influence of atorvastatin on salusin-alpha or associated with a decrease in serum lipid level; 3) salusin-alpha may predict mortality in HD patients.

DETAILED DESCRIPTION:
Purpose I, step 1. To investigate whether plasma salusin-alpha is associated with lipid and lipid-related abnormalities in hemodialysis (HD) patients, plasma salusin-alpha concentration, expression of receptor CD36 on macrophages, serum lipid parameters, anthropometric and laboratory indices of nutrition and biomarkers of inflammation will be cross-sectionally analyzed. In chronic kidney disease (CKD) patients there is a close association between atherosclerosis (A), malnutrition (M) and inflammation (I), known as MIA syndrome, so interactions between all these parameters will be obviously present and should be taken into account. In addition, homeostasis model assessment of insulin resistance (HOMA-IR) will be applied as insulin resistance is a metabolic abnormality occurring in advanced CKD, in metabolic syndrome shown in about 50% of HD patients and diabetic mellitus (DM), being a cause of CKD in approximately 40% of cases. Results of correlations and associations shown in HD patients will be compared with those of healthy controls and obese persons with normal renal function for evaluation of salusin-alpha relationships under different metabolic conditions, which may exert not uniform influence.

Study populations:

HD patients (n = 200) Obese persons (n = 50) Controls (n = 60)

Data collection:

Medical history (with special attention for demographics - age, gender, cause of CKD, renal replacement therapy vintage, changes in body weight, habits and data required for inclusion and exclusion criteria.

Physical examination (with special attention for skin abnormalities related to lipid disturbances and blood pressure).

Anthropometric indices:

* directly measured: height, body weight, hip and waist circumferences, midarm circumference (MAC), triceps skin fold thickness (TSF)
* calculated or estimated: hip to waist ratio (WHiR), height to waist ratio (WHeR), body mass index (BMI), in HD patients - dry body weight (DBW) Laboratory parameters
* Apolipoprotein A1 (APOA1)
* Apolipoprotein B (APO B)
* Cholesterol - total
* Cholesterol HDL
* Cholesterol LDL directly measured
* CD36
* Free fatty acids (FDA)
* High sensitivity C-reactive protein (hsCRP)
* HOMA-IR
* Interleukin 6 (IL-6)
* L-carnitine
* Lipase
* Lipoprotein(a)
* Salusin-alpha
* Triglycerides
* Basic serum biochemistry

Purpose I, step 2. HD patients suffering from type 2DM or having metabolic syndrome (MeS) are at risk of more severe lipid abnormalities than the remaining ones. Data collected in Step 1 will be helpful in diagnosis of MeS in the examined HD patients. The investigators expect that also in controls they will find persons with abnormal serum lipid profile. Differences inside these both groups may influence plasma salusin-alpha levels and the examined associations. Thereby, the following groups will be analyzed separately and compared to each other:

For HD patients:

* group with MeS and with type 2 DM
* group only with MeS
* group only with type 2 DM
* group without MeS and without DM

For controls:

* group without detected serum lipid abnormalities
* group with detected serum lipid abnormalities

Validation of correlations/associations found in the cross-sectional study will be done in the prospective studies (Purpose II) and at the final analysis (Purpose III).

Purpose II. The treatment with atorvastatin lowers serum LDL cholesterol in HD patients. Using this statin during the study, the investigators can observe dynamic changes in serum LDL cholesterol in HD patients with known plasma salusin-alpha concentration before atorvastatin medication. With repeated salusin-alpha measurements during continued atorvastatin treatment the investigators can follow concomitantly occurring (or not occurring) changes in plasma salusin-alpha concentrations, which can be related to atorvastatin directly or to its LDL cholesterol lowering effect. To elucidate this aspect, the investigators plan to examine hyperlipidemic HD patients treated with a prescribed diet and increased physical activity as well as obese persons (not taking lipid lowering medication) during weight lowering therapy, which usually decreases lipidemia. Results of these persons may give the answer whether a decrease in lipidemia without pharmaceutical medication leads (may be also leads) to changes in plasma salusin-alpha concentration.

The prospective study is planned in two groups of persons:

HD patients, participating in Step 1 (n = 200), Obese persons, participating in Step 1 (n = 50).

Purpose III. Annual mortality rate in HD patients is 10 - 15%. LDL cholesterol and total cholesterol are predictors of mortality in end-stage renal disease patients. If salusin-alpha is associated with lipid abnormalities, it is a reasonable to check whether this peptide may be a predictor of mortality in HD patients. To investigate this aspect the investigators plan to perform the analysis of HD patients outcome after two years from the first salusin-alpha determination and to check whether there is any association between plasma salusin-alpha concentration and death from cardiovascular events and all cause death.

ELIGIBILITY:
Inclusion Criteria:

For HD patients:

* HD vintage at least 3 months
* signed consent for participation in the study

For obese persons:

* BMI > 30 kg/m2
* eGFR > 60 ml/min/1.73 m2 BSA
* interest in weight loss according to weight loss diet protocol (WLDP)
* signed consent for participation in the study

For controls (healthy volunteers):

* declared health, comfort
* no substantial changes in the medical interview and physical examination
* no medication
* signed consent for participation in the study

Exclusion Criteria:

For HD patients:

* active thyroid gland disease and/or thyreotropic medication
* treatment with corticosteroids, immunosuppressants or hormones
* treatment with statins or fibrates in 6 weeks before the study commencement
* diagnosis of genetic lipid abnormalities
* neoplastic disease
* acute coronary syndrome and/or cerebral stroke in 6 months before the study commencement
* surgery in 3 months before the study commencement
* plasma activities of ALT and/or AST exceeding 3 times the upper laboratory normal limit
* non compensated diabetes mellitus

For obese persons:

* a known history of moderate or severe cardiovascular disease, stroke or transient ischemic attack
* uncontrolled hypertension
* severe dyslipidemia (triglycerides > 500 mg/dl, total cholesterol > 350 mg/dl) or taking lipid-lowering agents at the recruitment or 6 weeks before
* serious chronic disease requiring active treatment (example with glucocorticoids, antineoplastic agents, psychoactive agents, bronchodilators on a regular basis, insulin or oral hypoglycemic drugs)
* women of child-bearing potential using an effective form of hormonal birth control, pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2011-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
normalization of serum LDL cholesterol | 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alicja E. Grzegorzewska, MD, PhD, Study Chair — Chair and Department of Nephrology, Transplantology and Internal Diseases; Leszek Niepolski, MD, PhD, Principal Investigator — BBraun Avitum Dialysis Center
Locations (1):
- BBraun Avitum Dialysis Center, Nowy Tomyśl, Wielkopolska, Poland

REFERENCES:
- [Background] Watanabe T, Sato K, Itoh F, Iso Y, Nagashima M, Hirano T, Shichiri M. The roles of salusins in atherosclerosis and related cardiovascular diseases. J Am Soc Hypertens. 2011 Sep-Oct;5(5):359-65. doi: 10.1016/j.jash.2011.06.003. PMID 21925457
- [Background] Ti Y, Wang F, Wang ZH, Wang XL, Zhang W, Zhang Y, Bu PL. Associations of serum salusin-alpha levels with atherosclerosis and left ventricular diastolic dysfunction in essential hypertension. J Hum Hypertens. 2012 Oct;26(10):603-9. doi: 10.1038/jhh.2011.71. Epub 2011 Aug 11. PMID 21833023
- [Background] Suzuki N, Shichiri M, Tateno T, Sato K, Hirata Y. Distinct systemic distribution of salusin-alpha and salusin-beta in the rat. Peptides. 2011 Apr;32(4):805-10. doi: 10.1016/j.peptides.2010.12.012. Epub 2010 Dec 28. PMID 21193001
- [Background] Ozgen M, Koca SS, Dagli N, Balin M, Ustundag B, Isik A. Serum salusin-alpha level in rheumatoid arthritis. Regul Pept. 2011 Feb 25;167(1):125-8. doi: 10.1016/j.regpep.2010.12.003. Epub 2010 Dec 24. PMID 21185876
- [Background] Nagashima M, Watanabe T, Shiraishi Y, Morita R, Terasaki M, Arita S, Hongo S, Sato K, Shichiri M, Miyazaki A, Hirano T. Chronic infusion of salusin-alpha and -beta exerts opposite effects on atherosclerotic lesion development in apolipoprotein E-deficient mice. Atherosclerosis. 2010 Sep;212(1):70-7. doi: 10.1016/j.atherosclerosis.2010.04.027. Epub 2010 May 4. PMID 20684826